CLINICAL TRIAL: NCT00751946
Title: Girls In Recovery From Life Stress (GIRLS) Study
Acronym: GIRLS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: U.S. Department of Justice (U.S. Federal Agency)
Responsible Party: Julian Ford, Ph.D., University of Connecticut Health Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-035H-2; 2005-MU-MU-K013
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2010-09-27 (Estimated); Status verified 2010-09

CONDITIONS: Posttraumatic Stress Disorder; PTSD
Keywords: Posttraumatic Stress Disorder; PTSD; psychotherapy; adolescents; clinical trial
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 12 weekly sessions of one-to-one TARGET (psychotherapy)
  Interventions: Behavioral: Trauma Adaptive Recovery Group Education and Therapy
- 2 (Active Comparator): 12 weekly sessions of one-to-one ETAU (psychotherapy)
  Interventions: Behavioral: Enhanced Treatment As Usual

INTERVENTIONS:
Behavioral: Trauma Adaptive Recovery Group Education and Therapy — Trauma Affect Regulation: Guidelines for Education and Therapy (TARGET; Ford & Russo, 2006) is a manualized gender-specific treatment for PTSD. The 12-session individual therapy version in the present study is being adapted for adolescent girls based on a parallel version for young mothers and a group version that has been field tested with more than 20 adolescent girls.
  TARGET teaches a practical 7-step sequence of skills for processing and managing trauma-related reactions to current stressful experiences. The skills are designed in a sequence mirroring the three phases of complex traumatic stress disorder treatment (Ford, Courtois, Van der Hart, Nijenhuis & Steele, 2005), summarized by an acronym "FREEDOM". TARGET also uses creative arts activities: personalized "lifelines" via collage, drawing, poetry, and writing.
  Arms: 1
Behavioral: Enhanced Treatment As Usual — Enhanced Treatment as Usual (ETAU) is a 12-session supportive therapy adapted from the Present Centered Therapy co-developed by the first author (McDonagh-Coyle, Friedman, McHugo, Ford, Mueser, & Sengupta, 2005). In ETAU therapists invite the participant to talk about goals or problems that are important to her. The therapist's focus is on providing the core conditions of client centered psychotherapy (nonjudgmental acceptance, empathy, interpersonal warmth) and engaging the participant in a strengths-based solution-focused reflection on how she is successful (or has been in the past) in managing stressors, handling problems, achieving personal goals, and developing healthy relationships with peers, family, and other community members.
  Arms: 2

SUMMARY:
This study will compare treatment outcomes of 90 adolescent girls who are (a) at high risk for delinquency and/or are juvenile justice involved, and (b) who are experiencing symptoms of PTSD: 45 of the girls will receive Trauma Affect Regulation: Guide for Education and Therapy (TARGET, Frisman, Ford, Lin, Mallon, & Chang, in press), and their outcomes will be compared to 45 girls who receive Enhanced Treatment as Usual (ETAU). As part of their involvement, participants will make phone calls to provide data via an interactive voice response system (IVR), meet 3 times for a research interview, and be invited to participate in a cognitive assessment substudy at the Olin Neuropsychiatric Research Center at Hartford Hospital.

DETAILED DESCRIPTION:
Hypotheses, Objectives and Aims:

The purpose of the GIRLS study is to provide counseling to adolescent girls who are (a) at high risk for delinquency and/or are juvenile justice involved and (b) are experiencing symptoms of PTSD, in order to help them regulate their emotions, planning, decision-making, and actions/ interactions in ways that will reduce PTSD and enhance their safety, responsible civic involvement, learning, peer, family, and adult relationships, and physical and psychological well-being. The study will be the first randomized clinical trial of a therapeutic intervention for complex post-traumatic stress disorder (PTSD)with girls: 1) Trauma Affect Regulation: Guide for Education and Therapy (TARGET; Frisman, Ford, Lin, Mallon, & Chang, in press), compared to Enhanced Treatment as Usual (ETAU). Both interventions will provide 12 one-to-one manualized, educational and therapeutic sessions that teach coping skills and stress reduction techniques.

The aims of the study are:

Aim 1) To test if participation in TARGET results in clinically and statistically significant improvements in PTSD symptoms, psychosocial functioning, and emotion/impulse regulation.

Aim 2) To compare the differential affects of TARGET and ETAU on affect regulation, social support, stress-related information processing and cognitive coping, and the reduction of impulsive or aggressive thinking/behavior.

Aim 3) To identify changes in daily self-regulation after TARGET and ETAU.

An ethnically diverse sample of girls at high risk for delinquency and/or with current or past juvenile justice-involvement between 13 and 17 years of age will be recruited in clinic, community, detention, schools, and residential programs. After screening for eligibility and obtaining valid signed consent forms, participants will be randomly assigned to one of the two experimental conditions. Within each condition, trained clinicians will administer 12 sessions of individualized counseling using a manual for the intervention. Psychometric self-report and daily monitoring measures will be obtained at baseline, post-treatment, and 6-month follow-up assessments and multivariate statistical techniques will be used for analysis of treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 13-17 years old
* Past and/or current juvenile justice involvement AND/OR past and/or current delinquent behavior
* Able to obtain assent from youth
* Able to obtain consent from legal guardian
* Willing to assent/consent to be audiotaped for research purposes in assessment and intervention sessions
* Currently experiencing negative reactions to past traumas (PTSD symptoms)

Exclusion Criteria:

* Imminently suicidal
* Past 30 days inpatient psychiatric treatment
* IF meetings take place at a school or group facility and the girl/participant is NOT willing to schedule appointments through the school or group facility staff

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2006-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Interview (CAPS-CA) assessing posttraumatic stress disorder and questionnaires (PTCI, IPSI, TMQ, TSCC) and clinician ratings (SOTS) assessing posttraumatic stress symptom severity. | Post-treatment, 4-6 months post-treatment

SECONDARY OUTCOMES:
Questionnaires assessing problems with externalizing behaviors (Weinberger Adjustment Survey) and socioemotional strengths (Hope, NMR, Weinberger Adjustment Survey) | Post-treatment and 4-6 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Julian Ford, Ph.D., Principal Investigator — UConn Health; Kathie H Moffitt, Ph.D., Study Director — UConn Health
Locations (7):
- United States (7):
  - Polaris School, East Hartford, Connecticut
  - University of Connecticut Health Center, Farmington, Connecticut
  - Gray Lodge Shelter for Women, Hartford, Connecticut
  - Weaver High School, Hartford, Connecticut
  - Bellizzi Middle School, Hartford, Connecticut
  - Quirk Middle School, Hartford, Connecticut
  - UCONN Health Partners, West Hartford, Connecticut

REFERENCES:
- [Background] Ford JD, Courtois CA, Steele K, Hart Ov, Nijenhuis ER. Treatment of complex posttraumatic self-dysregulation. J Trauma Stress. 2005 Oct;18(5):437-47. doi: 10.1002/jts.20051. PMID 16281241
- [Background] Ford JD, Russo E. Trauma-focused, present-centered, emotional self-regulation approach to integrated treatment for posttraumatic stress and addiction: trauma adaptive recovery group education and therapy (TARGET). Am J Psychother. 2006;60(4):335-55. doi: 10.1176/appi.psychotherapy.2006.60.4.335. PMID 17340945
- [Background] Frisman, L., Ford, J. D., Lin, H., Mallon, S., & Chang, R. (in press). Outcomes of trauma treatment using the TARGET model. Journal of Groups in Addiction and Recovery.
- [Background] McDonagh A, Friedman M, McHugo G, Ford J, Sengupta A, Mueser K, Demment CC, Fournier D, Schnurr PP, Descamps M. Randomized trial of cognitive-behavioral therapy for chronic posttraumatic stress disorder in adult female survivors of childhood sexual abuse. J Consult Clin Psychol. 2005 Jun;73(3):515-24. doi: 10.1037/0022-006X.73.3.515. PMID 15982149